CLINICAL TRIAL: NCT00785538
Title: Phase I Study of Anti-Insulin-Like Growth Factor-I Receptor (IGF-IR) Monoclonal Antibody IMC-A12 in Patients With Advanced Solid Tumors Who No Longer Respond to Standard Therapy or for Whom No Standard Therapy is Available
Brief Title: A Study of IMC-A12 in Participants With Tumors Who No Longer Respond to Treatment or For Whom No Treatment is Available
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 13932; CP13-0501 (Other: ImClone, LLC); I5A-IE-JAEH (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Advanced Solid Tumors
Keywords: Tumors; Antibodies, Monoclonal
MeSH Terms: conditions — Neoplasms | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-A12 (Experimental): All participants will receive intravenous (I.V.) infusions of IMC-A12, with the dose depending on which cohort they are enrolled into. A minimum of three participants will be enrolled in each cohort. When all participants complete a cohort, dose escalation to the next cohort will occur.
  Interventions: Biological: IMC-A12

INTERVENTIONS:
Biological: IMC-A12 — Cohort 1
  3 milligrams/kilogram (mg/kg), I.V. once a week, for 4 weeks, followed by a 2-week observation period.
  Other Names: Cixutumumab; LY3012217
Biological: IMC-A12 — Cohort 2
  6 mg/kg, I.V. once a week, for 4 weeks, followed by a 2-week observation period.
  Other Names: Cixutumumab; LY3012217
Biological: IMC-A12 — Cohort 3
  10 mg/kg, I.V. once a week, for 4 weeks, followed by a 2-week observation period.
  Other Names: Cixutumumab; LY3012217
Biological: IMC-A12 — Cohort 4
  15 mg/kg, I.V. once a week, for 4 weeks, followed by a 2-week observation period.
  Other Names: Cixutumumab; LY3012217
Biological: IMC-A12 — Cohort 5
  21 mg/kg, I.V. once a week, for 4 weeks, followed by a 2-week observation period.
  Other Names: Cixutumumab; LY3012217
Biological: IMC-A12 — Cohort 6
  27 mg/kg, I.V. once a week, for 4 weeks, followed by a 2-week observation period.
  Other Names: Cixutumumab; LY3012217

SUMMARY:
The purpose of this study is to determine if IMC-A12 is safe for participants, and also to determine the best dose of IMC-A12 to give to participants.

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety profile and maximum tolerated dose (MTD) of the anti-IGF-IR monoclonal antibody IMC-A12 administered weekly in participants with advanced solid tumors who no longer respond to standard therapy or for whom no standard therapy is available

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically-documented, measurable, advanced primary or recurrent solid tumors that no longer respond to standard therapy or for which no standard therapy is available.
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2 at study entry
* Able to provide written informed consent
* Life expectancy of >3 months
* Adequate hematologic functions, as defined by: absolute neutrophil count (ANC) ≥1500/cubic millimeter (mm³), hemoglobin level ≥10 grams/deciliter (gm/dL), platelet count ≥100,000/mm³
* Adequate hepatic function, as defined by: total bilirubin level ≤1.5 x the upper limit of normal (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤2.5 x the ULN or ≤5 x the ULN if known liver metastases
* Adequate renal function, as defined by a serum creatinine level ≤1.5 x the ULN
* Ejection fraction within the normal institutional limits
* Use of effective contraception per institutional standard, if procreative potential exists
* At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, prior radiation therapy (palliative radiation therapy is allowed), an open biopsy, or a significant traumatic injury to allow for adequate recovery. Ongoing side effects due to these agents must be ≤Grade 2 prior to entering the study.
* At least 6 weeks must have elapsed from nitrosoureas, mitomycin C, or monoclonal antibody [not targeting the insulin-like growth factor receptor (IGFR)] therapy to allow for adequate recovery. Ongoing side effects due to these agents must be ≤Grade 2 prior to entering the study.
* Accessible for treatment and follow-up. Participants enrolled in this trial must be treated at the participating center.

Exclusion Criteria:

* Any concurrent malignancy other than non-melanomatous skin cancer or carcinoma in situ of the cervix. Participants with a previous malignancy but without evidence of disease for ≥3 years will be allowed to enter the trial.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, unstable angina pectoris, angioplasty, stenting or myocardial infarction within 6 months, uncontrolled hypertension, clinically significant cardiac arrhythmia, psychiatric illness/social situations that would compromise participant safety or limit compliance with study requirements, participants with symptomatic brain metastases
* Serious or nonhealing active wound, ulcer or bone fracture
* Know human immunodeficiency virus (HIV)-positive
* History of hemorrhagic or thrombotic disorder within 9 months
* Proteinuria ≥1+ by routine urinalysis (participants with a protein value of ≤500 milligrams (mg) confirmed by a 24-hour urine collection are eligible)
* Pregnant [confirmed by serum beta human chorionic gonadotropin (βHCG)] or breast feeding
* History of prior treatment with other agents specifically targeting IGFRs
* Known diabetes
* Inability or unwillingness to interrupt steroidal or hormonal therapy for the duration of treatment with IMC-A12
* Positive anti-IMC-A12 antibody response
* History of allergic reactions to monoclonal antibodies or other therapeutic proteins
* Employees of the investigator or study center with direct involvement in this study or other studies under the direction of the investigator or study center, as well as family members of the employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - ImClone Investigational Site, Scottsdale, Arizona
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Higano CS, Berlin J, Gordon M, LoRusso P, Tang S, Dontabhaktuni A, Schwartz JD, Cosaert J, Mehnert JM. Safety, tolerability, and pharmacokinetics of single and multiple doses of intravenous cixutumumab (IMC-A12), an inhibitor of the insulin-like growth factor-I receptor, administered weekly or every 2 weeks in patients with advanced solid tumors. Invest New Drugs. 2015 Apr;33(2):450-62. doi: 10.1007/s10637-015-0217-7. Epub 2015 Mar 7. PMID 25749986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For participants enrolled under Protocol Versions 1.0 and 2.0, there was a 2-week pharmacokinetic (PK) period prior to Cycle 1.
Pre-assignment Details: After completion of the 10 milligrams/kilogram (mg/kg) cohort, PK data were obtained that established a recommended dose for Phase 2 studies. Enrollment and dose escalation beyond 15 mg/kg was stopped. Participants with progressive disease (PD) or death were considered to have completed the study.
Groups:
- 3 mg/kg: 3 mg/kg IMC-A12 administered intravenously (I.V.) on Day 1 of a 2-week PK period prior to Cycle 1.
  3 mg/kg IMC-A12 administered I.V. once a week for 4 weeks, for a total of 4 doses per cycle. Cycle 1 was followed by a 2-week observation.
  Participants with an objective response after Cycle 1 could have received additional treatment cycles at the same dose and schedule until disease progression or withdrawal criteria were met. Participants with stable disease (SD) could have received up to 2 additional 4-week treatment cycles at the same dose and schedule.
- 6 mg/kg: 6 mg/kg IMC-A12 administered I.V. on Day 1 of a 2-week PK period prior to Cycle 1.
  6 mg/kg IMC-A12 administered I.V. once a week for 4 weeks, for a total of 4 doses per cycle. Cycle 1 was followed by a 2-week observation.
  Participants with an objective response after Cycle 1 could have received additional treatment cycles at the same dose and schedule until disease progression or withdrawal criteria were met. Participants with SD could have received up to 2 additional 4-week treatment cycles at the same dose and schedule.
- 10 mg/kg: 10 mg/kg IMC-A12 administered I.V. on Day 1 of a 2-week PK period prior to Cycle 1.
  10 mg/kg IMC-A12 administered I.V. once a week for 4 weeks, for a total of 4 doses per cycle. Cycle 1 was followed by a 2-week observation.
  Participants with an objective response after Cycle 1 could have received additional treatment cycles at the same dose and schedule until disease progression or withdrawal criteria were met. Participants with SD could have received up to 2 additional 4-week treatment cycles at the same dose and schedule.
- 15 mg/kg: 15 mg/kg IMC-A12 administered I.V. once a week for 4 weeks, for a total of 4 doses per cycle. Cycle 1 was followed by a 2-week observation.
  Participants with an objective response after Cycle 1 could have received additional treatment cycles at the same dose and schedule until disease progression or withdrawal criteria were met. Participants with SD could have received up to 2 additional 4-week treatment cycles at the same dose and schedule.
Period: PK Period
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Started | 7 | 1 | 1 | 0
Completed | 7 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Started | 7 | 9 | 6 | 2
Received at Least 1 Dose of Study Drug | 7 | 9 | 6 | 2
Completed | 6 | 7 | 4 | 1
Not Completed | 1 | 2 | 2 | 1
Not completed — Adverse Event | 1 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 3 mg/kg: 3 mg/kg IMC-A12 administered I.V. on Day 1 of a 2-week PK period prior to Cycle 1.
  3 mg/kg IMC-A12 administered I.V. once a week for 4 weeks, for a total of 4 doses per cycle. Cycle 1 was followed by a 2-week observation.
  Participants with an objective response after Cycle 1 could have received additional treatment cycles at the same dose and schedule until disease progression or withdrawal criteria were met. Participants with SD could have received up to 2 additional 4-week treatment cycles at the same dose and schedule.
- Total: Total of all reporting groups
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 6 | 2 | 24
Age, Continuous [Median (Full Range); unit: years] | 65.7 (10.43) [45 to 70] | 56.4 (6.30) [47 to 67] | 59.4 (15.17) [25 to 69] | 42.9 (15.13) [32 to 54] | 57.2 (11.13) [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 1 | 10
  Male | 4 | 4 | 5 | 1 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 8 | 5 | 1 | 18
  Black | 1 | 1 | 0 | 1 | 3
  Asian | 1 | 0 | 1 | 0 | 2
  Hispanic | 0 | 0 | 0 | 0 | 0
  Unknown | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 6 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) or Deaths
Description: Data presented are the number of participants who experienced serious adverse events (SAEs), other non-serious AEs and deaths during the study including the 30-day follow-up. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Enrollment to study completion up to 215 weeks
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 7 | 9 | 6 | 2
Participants
  SAEs | 2 | 3 | 2 | 0
  AEs | 7 | 8 | 6 | 2
  Death due to PD | 0 | 1 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the dose preceding the dose level at which 2 participants experienced a dose-limiting toxicity (DLT). A DLT was defined as any Grade 3 or 4 hematologic or nonhematologic toxicity based on Common Terminology Criteria for AE (CTCAE), excluding alopecia, which was considered by the investigator to be definitely, probably, or possibly related to IMC-A12.
Time Frame: 6 weeks
Population: All participants who received at least 1 dose of study drug and completed Cycle 1 and 2-week observation or discontinued treatment for an IMC-A12-related toxicity.
Measure: Number; unit: mg/kg
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 6 | 7 | 5 | 1
mg/kg | NA — MTD was not reached because <2 participants experiencing a DLT. | NA — MTD was not reached because <2 participants experiencing a DLT. | NA — MTD was not reached because <2 participants experiencing a DLT. | NA — MTD was not reached because of early stopping based on PK results.

3. Secondary Outcome: Maximum Concentration (Cmax) of IMC-A12 Following Multiple Doses
Time Frame: Predose, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours after the infusion of Cycle 1
Population: All participants who received study drug and had PK data available to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 4 | 3 | 1 | 1
micrograms/milliliter (µg/mL) | 292 (42) | 385 (51) | 734 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated. | 965 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

4. Secondary Outcome: Observed Serum Concentration of IMC-A12 at 168 Hour Post End of Infusion Following Multiple Doses
Time Frame: Predose, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours after the infusion of Cycle 1
Population: All participants who received study drug and had PK data available to calculate Cmin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 3 | 2 | 1 | 1
µg/mL | 74.8 (28) | 154 (NA) — 2 participants were analyzed; therefore arithmetic mean was calculated and geometric coefficient of variation was not calculated. | 226 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated. | 122 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

5. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve of IMC-A12 During One Dosing Interval (AUCτ) Following Multiple Doses
Time Frame: Predose, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours after the infusion of Cycle 1
Population: All participants who received study drug and had PK data available to calculate AUCτ.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg*h/mL
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 3 | 2 | 1 | 1
micrograms*hour/milliliter (µg*h/mL | 19800 (39) | 36350 (NA) — 2 participants were analyzed; therefore arithmetic mean was calculated and geometric coefficient of variation was not calculated. | 66700 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated. | 49300 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

6. Secondary Outcome: Half-Life (t1/2) of IMC-A12 Following Multiple Doses
Description: Half-Life (t1/2) is the time measured for the plasma concentration of the drug to decrease by one half. The analysis was not performed for the 6 mg/kg and 10 mg/kg dosing groups due to insufficient PK data.
Time Frame: Predose, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours after the infusion of Cycle 1
Population: All participants who received study drug and had PK data available to calculate t1/2. Zero participants were analyzed for the 6 mg/kg and 10 mg/kg dosing groups due to insufficient PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 2 | 0 | 0 | 1
days | 6.19 (NA) — 2 participants were analyzed; therefore arithmetic mean was calculated and geometric coefficient of variation was not calculated. |  |  | 6.17 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

7. Secondary Outcome: Clearance Rate of IMC-A12 at Steady State (CLss) Following Multiple Doses
Description: CLss is the volume of plasma (or blood) from which the drug is completely removed, or cleared, in a given time at steady-state.
Time Frame: Predose, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours after the infusion of Cycle 1
Population: All participants who received study drug and had PK data available to calculate CLss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 3 | 2 | 1 | 1
Liters/hour (L/h) | 0.0124 (40) | 0.0125 (NA) — 2 participants were analyzed; therefore arithmetic mean was calculated and geometric coefficient of variation was not calculated. | 0.0114 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated. | 0.0296 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

8. Secondary Outcome: Volume of Distribution of IMC-A12 at Steady State (Vss) Following Multiple Doses
Description: Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug at steady-state. The analysis was not performed for the 6 mg/kg and 10 mg/kg dosing groups due to insufficient PK data.
Time Frame: Predose, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 hours after the infusion of Cycle 1
Population: All participants who received study drug and had PK data available to calculate Vss. Zero participants were analyzed for the 6 mg/kg and 10 mg/kg dosing groups due to insufficient PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 2 | 0 | 0 | 1
Liters (L) | 2.88 (NA) — 2 participants were analyzed; therefore arithmetic mean was calculated and geometric coefficient of variation was not calculated. |  |  | 5.19 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

9. Secondary Outcome: Serum Anti-IMC-A12 Antibody Assessment (Immunogenicity)
Description: Analysis was not performed due to lack of available assay.
Time Frame: Before the last infusion of each treatment cycle
Population: Zero participants were analyzed due to lack of available assay.
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Best Overall Response
Description: Stable Disease (SD) is neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for progressive disease (PD). PR and PD were assessed by investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PR is ≥30% decrease in sum of longest diameter of target lesions. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion. Participants with a global deterioration of their health status requiring discontinuation of treatment without objective evidence of disease progression at that time were to be reported as "symptomatic deterioration"
Time Frame: Enrollment to study completion up to 215 weeks
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Number analyzed (Participants) | 7 | 9 | 6 | 2
Participants
  Stable Disease (SD) | 2 | 1 | 2 | 1
  Progressive Disease (PD) | 5 | 4 | 2 | 1
  Symptomatic Deterioration | 0 | 3 | 0 | 0
  Not Evaluable | 0 | 1 | 2 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 3 mg/kg | 6 mg/kg | 10 mg/kg | 15 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/9 | 2/6 | 0/2
Other Adverse Events (participants affected / at risk) | 7/7 | 8/9 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg/kg (N=7) | 6 mg/kg (N=9) | 10 mg/kg (N=6) | 15 mg/kg (N=2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 3 mg/kg (N=7) | 6 mg/kg (N=9) | 10 mg/kg (N=6) | 15 mg/kg (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISUAL DISTURBANCE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (3)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EARLY SATIETY (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 2 (3) | 5 (5) | 1 (2)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NODULE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
HEPATIC PAIN (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HELICOBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DENTAL EXAMINATION ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPUTUM ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
SENSORY DISTURBANCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0/4 (0) | 0/4 (0) | 0/5 (0) | 1/1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0/3 (0) | 0/5 (0) | 1/1 (1) | 0/1 (0)
BREATH SOUNDS DECREASED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CRACKLES LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.